CLINICAL TRIAL: NCT04208061
Title: A Phase 1, 2-Panel, Fixed-Sequence, Open-Label Single-Center Study to Assess the Effect of Single and Multiple Doses of Darunavir in Combination With Cobicistat or Ritonavir on the Pharmacokinetics of Single Dose Dabigatran Etexilate in Healthy Subjects
Brief Title: A Study of Darunavir in Combination With Cobicistat or Ritonavir, and Dabigatran Etexilate in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108697; 2019-003328-19 (EudraCT Number); TMC114FD1HTX1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Ritonavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Panel 1: Dabigatran etexilate +DRV/COBI (Experimental): Participants will receive Treatment A (single dose of Dabigatran etexilate orally) on Day 1 followed by Treatment B (single dose of Darunavir/ cobicistat [DRV/COBI] as fixed dose combination tablet orally and single dose of dabigatran etexilate) on Day 4 followed by Treatment C ([DRV/COBI] as fixed dose combination tablet orally once daily from Day 5 to Day 20 and single dose of dabigatran etexilate on Day 18).
  Interventions: Drug: Dabigatran Etexilate; Drug: DRV/COBI
- Panel 2: Dabigatran etexilate +DRV+rtv (Experimental): Participants will receive Treatment D (single dose of dabigatran etexilate orally) on Day 1 followed by Treatment E (single doses of Darunavir, and ritonavir [rtv], and single dose of dabigatran etexilate on Day 4), followed by Treatment F (DRV and rtv orally once daily from Day 5 to Day 20 and single dose of dabigatran etexilate on Day 18).
  Interventions: Drug: Dabigatran Etexilate; Drug: Ritonavir; Drug: Darunavir

INTERVENTIONS:
Drug: Dabigatran Etexilate — Participants will receive single dose of dabigatran etexilate orally.
Drug: DRV/COBI — Participants will receive oral tablet of fixed dose combination (FDC) containing darunavir (DRV)/ cobicistat (COBI).
  Other Names: REZOLSTA
  Arms: Panel 1: Dabigatran etexilate +DRV/COBI
Drug: Ritonavir — Participants will receive ritonavir orally.
  Arms: Panel 2: Dabigatran etexilate +DRV+rtv
Drug: Darunavir — Participants will receive Darunavir orally.
  Arms: Panel 2: Dabigatran etexilate +DRV+rtv

SUMMARY:
The purpose of this study is to evaluate effect of single and repeated doses of darunavir (DRV) in combination with cobicistat (DRV/COBI) and with ritonavir (DRV+rtv) on the pharmacokinetics of single dose dabigatran etexilate (measured in plasma as free and total dabigatran) when co-administered in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI) (weight in kilogram [kg]/height^2 in square meters [m^2] ) between 18.0 and 30.0 kg/m^2 (inclusive) and body weight not less than 50.0 kg
* Must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study
* A woman must have a negative highly sensitive serum beta human chorionic gonadotropin (beta hCG) pregnancy test at screening, on Day -1 (only if the test performed at screening was greater than [>] 4 days before dosing), and at the end of the study
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug
* Must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 days after receiving the last dose of study drug

Exclusion Criteria:

* Clinically significant abnormalities during physical examination, vital signs, or 12 lead - electrocardiogram (ECG) at screening as deemed appropriate by the investigator
* With any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* With a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Has donated blood or blood products or had substantial loss of blood (more than 500 milliliter [mL]) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Has received an investigational drug or used an investigational medical device within 60 days before the first intake of study drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Dabigatran Etexilate (Free and Total) | Up to Day 18
  Cmax is the maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of Last Quantifiable Concentration (AUC[0-last]) of Dabigatran Etexilate (Free and Total) | Up to Day 18
  AUC(0-last) is the Area under the curve (AUC) from time 0 to the time of last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinite Time (AUC0-infinity) of Dabigatran Etexilate (Free and Total) | Up to Day 18
  AUC(0-infinity) is defined as area under the plasma concentration-time curve from time zero to infinite time.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | From signing of the ICF up to end of study (up to 8 weeks)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] LaRoche JK, Lanier J, Alvarenga R, Collins M, Costelloe T, Chiau A, Whetherly H, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored in-human clinical trials: life cycle assessments of clinical trials spanning multiple phases and disease areas. BMJ Open. 2025 Feb 19;15(2):e085364. doi: 10.1136/bmjopen-2024-085364. PMID 39971605
- [Derived] LaRoche JK, Alvarenga R, Collins M, Costelloe T, De Soete W, Faludi J, Rens K. Climate footprint of industry-sponsored clinical research: an analysis of a phase-1 randomised clinical study and discussion of opportunities to reduce its impact. BMJ Open. 2024 Jan 11;14(1):e077129. doi: 10.1136/bmjopen-2023-077129. PMID 38216192